CLINICAL TRIAL: NCT05611047
Title: Multicentre Randomized Blinded Controlled Study of Specific Telerehabilitation of Multidomain Cognitive Impairment in Multiple Sclerosis Using Mixed Evaluation and Ecological Validity
Brief Title: Telerehabilitation of Multidomain Cognitive Impairment in Multiple Sclerosis
Acronym: TELECOG-MS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: withdrawal of Celgene
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CHUBX 2021/60
Record Dates: First submitted 2022-08-30; First posted 2022-11-09 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Multiple Sclerosis
Keywords: Autoimmune Diseases of the Nervous System; Demyelinating Autoimmune Diseases; Demyelinating Diseases; Immune System Diseases; Nervous System Diseases; Pathologic Processes; cognitive impairment; ecological assessment; telerehabilitation
MeSH Terms: conditions — Multiple Sclerosis; Autoimmune Diseases of the Nervous System; Demyelinating Diseases; Immune System Diseases; Nervous System Diseases; Pathologic Processes; Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active cognitive rehabilitation (Experimental)
  Interventions: Other: Clinical assessment; Other: Classical cognitive evaluation of several domains:; Other: Ecological evaluation; Behavioral: Patent reported outcomes (PRO's); Other: Telerehabilitation : active procedure
- Sham cognitive rehabilitation (Active Comparator)
  Interventions: Other: Clinical assessment; Other: Classical cognitive evaluation of several domains:; Other: Ecological evaluation; Behavioral: Patent reported outcomes (PRO's); Other: Telerehabilitation : comparator procedure

INTERVENTIONS:
Other: Clinical assessment — MS history and MS treatments and Expanded Disability Status Scale (EDSS) score will be recorded
Other: Classical cognitive evaluation of several domains: — Information processing speed (IPS) Working memory (WM) Executive functions (EF) Episodic memory (EM) Premorbid intelligence quotient (IQ) Multidomain or complex task
Other: Ecological evaluation — Virtual reality task : Urban DailyCog©
Behavioral: Patent reported outcomes (PRO's) — Patent reported outcomes (PRO's) : Beck Depression Inventory (BDI), European Quality of Life-5 Dimensions (EQ-5D-5L) for Health-Related Quality of Life (HRQOL), Multiple Sclerosis Impact Scale-29 Items (MSIS-29), French version of the Modified Fatigue Impact Scale (EMISEP) and State trait anxiety inventory (STAI).
  Subjective cognitive deficits: Perceived Deficits Questionnaire (PDQ) and Cognitive Activities Questionnaire (DCAQ)
Other: Telerehabilitation : active procedure — The Cognitive rehabilitation (CR) consists of weekly 45 minutes online individual session with the unblinded Speech Therapist.
  Arms: Active cognitive rehabilitation
Other: Telerehabilitation : comparator procedure — Once per week over a 12-week period completed by daily online exercises performed by the patient 4 days a week.
  Arms: Sham cognitive rehabilitation

SUMMARY:
Treating cognitive impairment (CI) in multiple sclerosis (MS), the leading cause of disability due to nontraumatic neurological disease in young adults, is an important challenge. The contribution of CI to disability in MS has been increasingly recognized, and CI has been shown to decrease health-related quality of life (HR-QOL), even in the early stages of the disease. CI negatively impacts daily activities such as driving, vocational status, absenteeism, and instrumental activities in persons living with MS (PwMS). No medication has proven to have a consistent symptomatic effect on CI in MS, and disease-modifying therapies only have a small impact on CI progression.

CI in MS is dominated by a slowdown in information processing speed (IPS), as well as by disturbances of more specific cognitive functions such as attention, episodic memory (EM), working memory (WM) and executive function (EF). The alteration of IPS has consequences for WM, attention, EF and EM. IPS impairment predicts subsequent disability and vocational status and changes in quality of life (QOL).

Cognitive rehabilitation (CR) is the most promising approach for treating MS-related CI, as concluded by recent reviews and meta-analyses, despite important methodological shortcomings. Methodological limitations in early studies have led to disappointing results, and well-designed studies are still scarce. As noted recently, many studies lack a randomized controlled design that includes passive or active control conditions, primary neuropsychological end-points identified a priori, evidence of the sustainability of CR and the inclusion of near and far transfer outcomes. Tertiary outcomes of QOL, metacognition, or other patient-reported outcomes (PROs) are rarely used.

In view of the results of these different studies, the investigators propose a single-blind randomized controlled trial of a telerehabilitation program for MS associated CI, based on Rehacom software, using appropriates modules according to specific CI, but complemented by individual remote online rehabilitation sessions allowing a better adaptation of the program to the patient's deficit, a more efficient supervision and meta-cognitive work. This program will be evaluated in terms of effectiveness on neuropsychological tests, effectiveness on specific cognitive domains re-educated according to the impairments detected in the baseline, an ecological evaluation and the impact on daily cognitive functioning. Specific active rehabilitation will be compared to a placebo intervention of the same duration and intensity. Only a multi-center study will make it possible to achieve sufficient number of patients to meet these objectives.

ELIGIBILITY:
Inclusion Criteria:

* Male or female;
* Age 18-55 years;
* Native French speaking;
* Definite diagnosis of Relapsing-remitting MS (RRMS) according to McDonald 2017 criteria;
* Disease duration> 12 months and ≤ 15 years;
* Computerized-Screening Cognitive Test (CSCT) score ≤ - 1.282 Standard Deviations (SD) (10th percentile) and/or cognitive complaint;
* 3 scores -1 SDa or 2 scores -1.5 SDb at least 2 of 5 baseline preselection neuropsychological battery tests in one of the following domains: processing speed or attention or working memory (SDMT, subtests alert, divided attention, visual scanning for selective attention, TAP and subtest working memory of the WAIS IV) and SDMT score not ≤ -3 SD;
* Able to use a computer with Windows operating system, an internet connection;
* Being affiliated to health insurance
* Having signed an informed consent (at the latest on the day of inclusion and before any examination required by research)

Exclusion Criteria:

* Previous history of other neurological disease;
* Psychiatric comorbidity including severe depression according to Diagnostic and Statistical Manual-IV (DSM-IV);
* Current dependence on alcohol or other addiction to toxic;
* Disabling visual or motor problems preventing participation to neuropsychological assessments;
* Change of psychotropic drug or disease-modifying therapies since less than one month;
* MS relapse in the month preceding the inclusion visit
* Illiteracy, ie: unable to count or to read;
* Acquisition disorders: dyslexia, dysphasia, dyscalculia and dyspraxia;
* Pregnant or breastfeeding women;
* Patient concerned by articles L 1121-5 to L 1121-8 (persons deprived of their liberty by a judicial or administrative decision, minors, persons of legal age who are the object of a legal protection measure or unable to express their consent).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-02-21 (Actual); Primary Completion 2025-02-19 (Actual); Study Completion 2025-02-19 (Actual)

PRIMARY OUTCOMES:
Improvement of two of the four reaction time z scores over the 12 weeks of training in the ecological assessment of cognitive impairment (CI) using the Urban DailyCog®. | 12 weeks after baseline (Day 0)

SECONDARY OUTCOMES:
Change in the neuropsychological tests raw scores between baseline (W0) and after rehabilitation (W12) between the two groups | 12 weeks after baseline (Day 0)
Change in the neuropsychological tests raw scores between visit W12 and visit W24 between the two groups. | 24 weeks after baseline (Day 0)
Change in information processing speed (IPS), composite z scores between W0-W12 and W12-W24 | 24 weeks after baseline (Day 0)
Change in attention and working memory (WM) domain neuropsychological tests composite z scores and raw scores between W0-W12 and W12-W24 in subgroups of patients affected for these domains | 24 weeks after baseline (Day 0)
Change in the sum of the 4 reaction time differences over the 12 weeks of training in the ecological assessment of CI using the Urban DailyCog®. | 12 weeks after baseline (Day 0)
Change in the patient-reported outcomes (PROs) (depression anxiety) and Subjective cognitive deficits questionnaire (PDQ and DCAQ) between baseline (W0) and after rehabilitation (W12) between the two groups. | 12 weeks after baseline (Day 0)
Change in the patient-reported outcomes (PROs) (daily cognitive functioning) and Subjective cognitive deficits questionnaire (PDQ and DCAQ) between baseline (W0) and after rehabilitation (W12) between the two groups. | 12 weeks after baseline (Day 0)
Change in the patient-reported outcomes (PROs) (fatigue) and Subjective cognitive deficits questionnaire (PDQ and DCAQ) between baseline (W0) and after rehabilitation (W12) between the two groups. | 12 weeks after baseline (Day 0)
Change in the patient-reported outcomes (PROs) (Health-Related Quality of Life) and Subjective cognitive deficits questionnaire (PDQ and DCAQ) between baseline (W0) and after rehabilitation (W12) between the two groups. | 12 weeks after baseline (Day 0)
Change in the PROs (depression anxiety) and Subjective cognitive deficits questionnaire (PDQ and DCAQ) between W0 and the 24-weeks follow-up (W24) between the two groups. | 24 weeks after baseline (Day 0)
Change in the PROs (daily cognitive) and Subjective cognitive deficits questionnaire (PDQ and DCAQ) between W0 and the 24-weeks follow-up (W24) between the two groups. | 24 weeks after baseline (Day 0)
Change in the PROs (fatigue) and Subjective cognitive deficits questionnaire (PDQ and DCAQ) between W0 and the 24-weeks follow-up (W24) between the two groups. | 24 weeks after baseline (Day 0)
Change in the PROs (Health-Related Quality of Life) and Subjective cognitive deficits questionnaire (PDQ and DCAQ) between W0 and the 24-weeks follow-up (W24) between the two groups. | 24 weeks after baseline (Day 0)

CONTACTS AND LOCATIONS:
Overall Officials: Aurélie RUET, Prof, Principal Investigator — University Hospital, Bordeaux
Locations (7):
- France (7):
  - CHU de Bordeaux - Service de neurologie, Bordeaux
  - CHU de Clermont-Ferrand - Service de neurologie, Clermont-Ferrand
  - CHU de Dijon-Bourgogne - Service de neurologie, Dijon
  - CH de Dunkerque - Service de neurologie, Dunkirk
  - Hôpital Saint Vincent de Paul - Service de neurologie, Lille
  - CHU de Montpellier - Service de neurologie, Montpellier
  - CHI Hôpital de Poissy Saint Germain en Laye - Service de neurologie, Poissy

IPD SHARING:
Plan to Share IPD: No